CLINICAL TRIAL: NCT04408053
Title: Mini-invasive Preventive Fixation of the Contralateral Femoral Neck in Patients Operated on for a Femoral Neck Fracture
Acronym: PREFIX
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APHP180585
Record Dates: First submitted 2020-05-26; First posted 2020-05-29 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Femoral Neck Fractures
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preventive fixation of the contralateral femoral neck (Experimental): Mini-invasive preventive fixation of the contralateral femoral neck : 6.5mm titanium cannulated self-tapping/self-drilling screws (Stryker Trauma and Depuy Synthes) : 2 screws per patients
  Interventions: Device: Preventive fixation of the contralateral femoral neck (Stryker Trauma and Depuy Synthes screws)
- No fixation (No Intervention)

INTERVENTIONS:
Device: Preventive fixation of the contralateral femoral neck (Stryker Trauma and Depuy Synthes screws) — 6.5mm titanium cannulated self-tapping/self-drilling screws (Stryker Trauma and Depuy Synthes) : 2 screws per patients
  Arms: Preventive fixation of the contralateral femoral neck

SUMMARY:
In France, the annual incidence of hip fracture is about 80 000 with more than 75% of these fractures occurring in patients aged 80 years old or more. About 10% percent of patients presenting with a hip fracture will sustain a contralateral hip fracture, most within 3 years. The consequences of a hip fracture are dramatic: 20% of patients die in the first year and less than half those who survive regain their previous level of function. Hip fractures are invariably associated with chronic pain, reduced mobility, disability, and an increasing degree of dependence. The efficacy of pharmacological treatments to prevent a contralateral hip fracture is marginal and postponed and compliance is known to be poor.

Osteoporosis is associated with cortical thinning and trabecular bone loss. Therefore, the mini-invasive preventive fixation (MIPF) of the contralateral femoral neck is appealing. The effect is immediate and compliance is certain. Morbidity is minimal because it is performed during the same operation as the fixation of the femoral neck fracture.

The main objective of this study is to determine whether the mini-invasive preventive fixation (MIPF) of the contralateral femoral neck in patients having a femoral neck fracture is superior to no fixation regarding the occurrence of a contralateral hip fracture within 3 years.

ELIGIBILITY:
Inclusion Criteria:

* women and men
* 80 years or older
* operated on for a femoral neck fracture
* presenting one, or more, added clinical risk factor of hip fracture*
* a fragility fracture in the past five years
* a history of fall in the past 12 months (not considering the fall that led to the present fracture)
* a very high risk of falling: use of psychoactive medication or impaired vision or impaired neuromuscular function
* BMI lower than 20kg/m2
* giving her/his consent.
* affiliated to the social security

Exclusion Criteria:

* history of a contralateral proximal femoral fracture
* history of a surgical operation of the contralateral proximal femur
* ongoing infection (bone or soft-tissue) on the contralateral hip
* contraindication of MIPF of the contralateral hip
* non ambulatory patients
* patients already included in the study
* patients with contraindication to the medical devices under evaluation
* patients not suitable for a surgical procedure (including not suitable for an anaesthetic)
* patients with a benign or malignant bone lesion of the contralateral femur
* patients included in another clinical research which could directly have an effect on the femoral neck bone strength
* patients presenting with a grade 4 Kellgren-Lawrence osteoarthritis of the contralateral hip and reporting significant clinical symptoms
* patients with an life expectancy of less than 3 months
* patients with a legal representative (tutorship or guardianship) and insane patients will be excluded

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 812 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of a contralateral fracture of the proximal femur | at 3 years after randomization

SECONDARY OUTCOMES:
Mortality | within 3 years after randomization
Proportion of patients requiring surgery on the contralateral proximal femur regardless the reason | within 3 years after randomization
Patient's autonomy | at 3 months after randomization
  Patient's autonomy will be assessed using the AGGIR scale. The AGGIR scale has 10 physical and mental variables and seven variables relating to domestic and social activities; the former are discriminative and the latter illustrative variables. The rating depends on the person doing the activity on her/his own; however, material and technical aids are allowed (glasses, wheelchair, etc). Each variable can take one of three modalities: A (perform alone), C (cannot perform alone), and B (can perform alone but on conditions).
Patient's autonomy | at 1 year after randomization
  Patient's autonomy will be assessed using the AGGIR scale. The AGGIR scale has 10 physical and mental variables and seven variables relating to domestic and social activities; the former are discriminative and the latter illustrative variables. The rating depends on the person doing the activity on her/his own; however, material and technical aids are allowed (glasses, wheelchair, etc). Each variable can take one of three modalities: A (perform alone), C (cannot perform alone), and B (can perform alone but on conditions).
Patient's autonomy | at 2 years after randomization
  Patient's autonomy will be assessed using the AGGIR scale. The AGGIR scale has 10 physical and mental variables and seven variables relating to domestic and social activities; the former are discriminative and the latter illustrative variables. The rating depends on the person doing the activity on her/his own; however, material and technical aids are allowed (glasses, wheelchair, etc). Each variable can take one of three modalities: A (perform alone), C (cannot perform alone), and B (can perform alone but on conditions).
Patient's autonomy | at 3 years after randomization
  Patient's autonomy will be assessed using the AGGIR scale. The AGGIR scale has 10 physical and mental variables and seven variables relating to domestic and social activities; the former are discriminative and the latter illustrative variables. The rating depends on the person doing the activity on her/his own; however, material and technical aids are allowed (glasses, wheelchair, etc). Each variable can take one of three modalities: A (perform alone), C (cannot perform alone), and B (can perform alone but on conditions).
Patient's function | at 3 months after randomization
  Patient's function will be assessed using the Parker score. The Parker scale assessment of mobility rates three questions: able to get about the house; able to get out of the house; able to go shopping. Each question may be answered as "no difficulty", with an aid"; "with the help from another person"; "not at all". Answer are weighted from 3 (no difficulty) to 0 (not at all). The maximum mobility score is 9; the lowest is 0.
Patient's function | at 1 year after randomization
  Patient's function will be assessed using the Parker score. The Parker scale assessment of mobility rates three questions: able to get about the house; able to get out of the house; able to go shopping. Each question may be answered as "no difficulty", with an aid"; "with the help from another person"; "not at all". Answer are weighted from 3 (no difficulty) to 0 (not at all). The maximum mobility score is 9; the lowest is 0.
Patient's function | at 2 years after randomization
  Patient's function will be assessed using the Parker score. The Parker scale assessment of mobility rates three questions: able to get about the house; able to get out of the house; able to go shopping. Each question may be answered as "no difficulty", with an aid"; "with the help from another person"; "not at all". Answer are weighted from 3 (no difficulty) to 0 (not at all). The maximum mobility score is 9; the lowest is 0.
Patient's function | at 3 years after randomization
  Patient's function will be assessed using the Parker score. The Parker scale assessment of mobility rates three questions: able to get about the house; able to get out of the house; able to go shopping. Each question may be answered as "no difficulty", with an aid"; "with the help from another person"; "not at all". Answer are weighted from 3 (no difficulty) to 0 (not at all). The maximum mobility score is 9; the lowest is 0.
Proportion of patients receiving an antiosteoporotic treatment | at 3 months after randomization
Number of falls since the last follow-up visit | at 3 months after randomization
Number of falls since the last follow-up visit | at 1 year after randomization
Number of falls since the last follow-up visit | at 2 years after randomization
Number of falls since the last follow-up visit | at 3 years after randomization
Pain on the contralateral hip | at 3 months after randomization
  Patients will be asked to rate the level of pain of the contralateral hip using a visual analogic scale, which goes from 0 (no pain) to 10 (maximum pain imaginable).
Pain on the contralateral hip | at 1 year after randomization
  Patients will be asked to rate the level of pain of the contralateral hip using a visual analogic scale,, which goes from 0 (no pain) to 10 (maximum pain imaginable).
Pain on the contralateral hip | at 2 years after randomization
  Patients will be asked to rate the level of pain of the contralateral hip using a visual analogic scale,, which goes from 0 (no pain) to 10 (maximum pain imaginable).
Pain on the contralateral hip | at 3 years after randomization
  Patients will be asked to rate the level of pain of the contralateral hip using a visual analogic scale,, which goes from 0 (no pain) to 10 (maximum pain imaginable).

IPD SHARING:
Plan to Share IPD: Undecided